CLINICAL TRIAL: NCT03923361
Title: Neural and Antidepressant Effects of Propofol (Phase 2)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in study design based on phase 1 data collection; patient burden was not feasible
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00116093B
Record Dates: First submitted 2019-04-19; First posted 2019-04-22 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propofol (Experimental)
  Interventions: Drug: Diprivan

INTERVENTIONS:
Drug: Diprivan — Similar to the high-intensity propofol treatments in Phase 1, the anesthesiologist will administer an induction dose of propofol followed by a continuous infusion, insert an airway, and begin mechanical ventilation. Propofol dosing will be adjusted with the goal of achieving a burst-suppression state with a SR of 40-60 for 12-15 minutes.
  Other Names: Propofol

SUMMARY:
Moderate-intensity propofol treatments will be administered to participants who are non-responders at the end of Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Diagnosis of major depressive disorder or bipolar disorder
* Current moderate-to-severe depressive episode
* Episode duration more than 2 months and less than 5 years
* Failure of at least 2 adequate antidepressant medication trials within the past 2 years
* Body mass index < 40
* 16-item Quick Inventory of Depressive Symptomatology, self-rated > 10

Exclusion Criteria:

* Contraindication to propofol or midazolam
* Daily use of benzodiazepine, opioid, ACE inhibitor, or ARB medication
* Symptomatic coronary artery disease or heart failure
* Poorly controlled hypertension or diabetes
* Abnormal kidney or liver function
* Pregnant or breast feeding
* Traumatic brain injury or significant neurologic signs (past year)
* Substance use disorder (past year)
* Obsessive compulsive disorder (current)
* Post-traumatic stress disorder (current)
* Schizophrenia-spectrum disorder (lifetime)
* Neurocognitive disorder (current)
* Personality disorder as a current focus of treatment
* ECT within the past 3 months
* Inappropriate for ECT, or poor response to ECT within the past 5 years
* Incompetent to provide consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 3 weeks after baseline
  24-item Hamilton Depression Rating Scale, total score Higher values represent more severe depressive symptoms Maximum score, 76; minimum score, 0 Remission defined as total score < 10 Response defined as decrease of total score from baseline > 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy Neuropsychiatric Institute, Salt Lake City, Utah, United States